CLINICAL TRIAL: NCT01920308
Title: A Prospective Study of the Performance of the Bard® LifeStent® Vascular Stent Systems (REALITY)
Acronym: REALITY
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BPV-13-001
Record Dates: First submitted 2013-08-08; First posted 2013-08-09 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 5 mm Bard LifeStent Vascular Stent: The study population will be comprised of subjects who present with moderate lifestyle-limiting claudication to mild tissue loss (Rutherford Category 2-5) that are candidates for PTA and stenting.
  Subjects with lesion(s) in the infra-inguinal segment (SFA and/or popliteal artery) will be considered for enrollment. The reference vessel diameter will be appropriate for treatment with available stent diameter of 5.0 mm (by visual estimate).
  Interventions: Device: 5 mm Bard LifeStent Vascular Stent

INTERVENTIONS:
Device: 5 mm Bard LifeStent Vascular Stent — The LifeStent® Vascular Stent is a peripheral stent intended to improve luminal diameter in the treatment of symptomatic de-novo or restenotic lesions up to 240 mm in length in the native superficial femoral artery (SFA) and popliteal artery with reference vessel diameters ranging from 4.0 - 6.5 mm.
  Other Names: Bard LifeStent Vascular Stent System; SFA stenting

SUMMARY:
The purpose of this study is to assess the deliverability, clinical utility and effectiveness of the 5 mm diameter size offering of the LifeStent® Vascular Stent

ELIGIBILITY:
Inclusion Criteria:

* The subject or legal representative has been informed of the nature of the evaluation, agrees to its provisions, and has signed the informed consent form (ICF)
* Subject agrees to comply with the protocol-mandated follow-up procedures and visits
* The subject is ≥ 21 years old
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within seven days prior to index procedure. Female subjects who are surgically sterile or post-menopausal are exempt from having a pregnancy test
* The subject has moderate lifestyle-limiting claudication to mild tissue loss defined as: Rutherford Category1 2-5 (moderate claudication to minor tissue loss
* The target lesion(s) has angiographic evidence of stenosis or restenosis ≥50% or occlusion in the SFA and/or popliteal artery (by visual estimate) and is amenable to PTA and stenting
* The target vessel reference diameter will be (by visual estimate) appropriate for treatment with available stent diameter of 5.0 mm
* A total of two stents may be used to cover lesions. Overlapping is allowed
* There is angiographic evidence of at least one vessel runoff to the foot (at the level of the malleolus

Exclusion Criteria:

* The subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with the study follow-up procedure and visits
* The subject has claudication or critical limb ischemia described as Rutherford Category1 0 (asymptomatic), 1 ( mild claudication), or 6 (major tissue loss)
* The subject has a known contraindication (including allergic reaction) or sensitivity to antiplatelet/anticoagulant medications, nickel, titanium or tantalum
* The subject has a known sensitivity to contrast media that is not amenable to pretreatment with steroids or/and antihistamines
* The subject has a history of bleeding diatheses or coagulopathy
* The subject has concomitant renal failure with a creatinine of >2.5 mg/dL
* The subject has concomitant hepatic insufficiency, thrombophlebitis, uremia, systemic lupus erythematosus (SLE), or deep vein thrombosis (DVT) at the time of the study procedure
* The subject is receiving dialysis or immunosuppressive therapy
* The subject is participating in an investigational drug or another investigational device study
* The subject has another medical condition, which, in the opinion of the investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with limited life expectancy of less than two years
* The subject has extensive peripheral vascular disease, which, in the opinion of the investigator, precludes safe insertion of an introducer sheath
* The target lesion(s) is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion(s)
* The subject has angiographic evidence of poor inflow, which would be deemed inadequate to support a vascular bypass graft
* The subject is diagnosed with septicemia at the time of the study procedure
* Patients with a stent previously implanted into the target vessel
* Lesions requiring the use of more than two stents
* Bilateral disease in the native SFA and/or proximal popliteal artery where both limbs meet the inclusion/exclusion criteria and it is planned to treat both limbs within 30 days. Note: One limb may be enrolled in the study, but only if the second limb is planned to be treated after the 30 day follow-up telephone screening has taken place. The limb that may be enrolled has to be the limb with the more severe lesion and the reasons for treating this specific limb will need to be stated in the CRF

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective observational study of the Bard® LifeStent® Vascular Stents in the treatment of symptomatic de novo or restenotic lesions.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Freedom from occurrence of death, amputation and TLR/TVR at 30 days post-index procedure. | 30 days
  30 day data can be collected via telephone screening. TLR is defined as a revascularization procedure (e.g. PTA (percutaneous transluminal angioplasty), cryoplasty, etc.) of the target lesion. TVR is defined as a revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) of the target vessel outside the target lesion.
Technical success, defined as successful deployment and placement accuracy based upon a rating scale completed by the investigators at time of index procedure. Book-end sizes will be evaluated for clinical utility of size range. | 30 days

SECONDARY OUTCOMES:
Secondary Safety defined as freedom from death (after 30 days) | Through 12 months post procedure
  Secondary Safety defined as freedom from death (after 30 days), stroke, MI, emergent surgical revascularization, significant distal embolization in target limb, target limb major amputation, and thrombosis of target vessel at 12 months post-index procedure.
Freedom from Target Lesion Revascularization (TLR) and/or Target Vessel Revascularization (TVR) after 30 days and 12 months post-index procedure. | Through 12 months
  TLR is defined as a revascularization procedure (e.g. PTA, cryoplasty, etc.) of the target lesion. TVR is defined as a revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) of the target vessel outside the target lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof. Dr., Principal Investigator — University Heart Centre in Bad Krozingen
Locations (1):
- University Heart Centre Bad Krozingen, Bad Krozingen, Germany